CLINICAL TRIAL: NCT02245555
Title: Observational Study About the Use of Tamsulosin in Patients With Benign Prostatic Hyperplasia
Brief Title: Observational Study of Tamsulosin in Patients With Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.73
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with benign prostatic hyperplasia
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: Secotex®

SUMMARY:
Study to describe Tamsulosin prescription characteristics in a representative population of patients on treatment for benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21 years old diagnosed with benign prostatic hyperplasia (BPH), who require pharmacological treatment to relieve symptoms and improve their quality of life, according to physician's judgment. The study will include naïve patients and patients not responding to previous therapy who receive Secotex as alternative or complementary treatment. The decision to treat a patient with Tamsulosin must be based on the best standard accepted in the clinical practice and must be carried out following Secotex (Tamsulosin) prescription information

Exclusion Criteria:

* Patients with known hypersensitivity to Tamsulosin or any of its ingredients, history of orthostatic hypotension or severe liver failure, or with any missing data required to complete the questionnaire are excluded

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign prostatic hyperplasia (BPH), who require pharmacological treatment
Sampling Method: Non-Probability Sample
Enrollment: 1060 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 21 months